CLINICAL TRIAL: NCT01725139
Title: A Randomised, Placebo-controlled, Double-blind, Repeat Dose Escalation Study With GSK2126458 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Proof of Mechanism Study With GSK2126458 in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 116711; 2012-001376-11 (EudraCT Number)
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — omipalisib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Cohort 1-GSK2126458 (Experimental): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 (0.25 mg twice daily [bid]) or placebo for approximately 8 days (7 to 10 days dosing)
  Interventions: Drug: GSK2126458
- Cohort 1-Placebo (Placebo Comparator): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or matching placebo for approximately 8 days (7 to 10 days dosing)
  Interventions: Drug: Placebo
- Cohort 2-GSK2126458 (Experimental): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or placebo for approximately 8 days (7 to 10 days dosing). GSK2126458 dose will be decided from Cohort 1 and which could be escalated or deescalated or repeated from Cohort 1 dosing.
  Interventions: Drug: GSK2126458
- Cohort 2-Placebo (Placebo Comparator): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or matching placebo for approximately 8 days (7 to 10 days dosing).
  Interventions: Drug: Placebo
- Cohort 3- GSK2126458 (Experimental): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or placebo for approximately 8 days (7 to 10 days dosing). GSK2126458 dose will be decided from Cohort 2 and which could be escalated or deescalated or repeated from Cohort 2 dosing.
  Interventions: Drug: GSK2126458
- Cohort 3-Placebo (Placebo Comparator): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or matching placebo for approximately 8 days (7 to 10 days dosing).
  Interventions: Drug: Placebo
- Cohort 4- GSK2126458 (Experimental): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or placebo for approximately 8 days (7 to 10 days dosing). GSK2126458 dose will be decided from Cohort 3 and which could be escalated or deescalated or repeated from Cohort 3 dosing.
  Interventions: Drug: GSK2126458
- Cohort 4- Placebo (Placebo Comparator): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or matching placebo for approximately 8 days (7 to 10 days dosing).
  Interventions: Drug: Placebo
- Cohort 5- GSK2126458 (Experimental): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or placebo for approximately 8 days (7 to 10 days dosing). GSK2126458 dose will be decided from Cohort 4 and which could be escalated or deescalated or repeated from Cohort 4 dosing.
  Interventions: Drug: GSK2126458
- Cohort 5- Placebo (Placebo Comparator): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or matching placebo for approximately 8 days (7 to 10 days dosing).
  Interventions: Drug: Placebo
- Cohort 6- GSK2126458 (Experimental): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or placebo for approximately 8 days (7 to 10 days dosing). GSK2126458 dose will be decided from Cohort 4 and which could be escalated or deescalated or repeated from Cohort 5 dosing.
  Interventions: Drug: GSK2126458
- Cohort 6- Placebo (Placebo Comparator): Subjects will be randomized in 3:1 ratio to receive either GSK2126458 bid or matching placebo for approximately 8 days (7 to 10 days dosing).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2126458 — GSK2126458 will be available as film coated tablet of dose strength 0.25 mg and 0.5 mg
  Arms: Cohort 1-GSK2126458; Cohort 2-GSK2126458; Cohort 3- GSK2126458; Cohort 4- GSK2126458; Cohort 5- GSK2126458; Cohort 6- GSK2126458
Drug: Placebo — Matching placebo will be available
  Arms: Cohort 1-Placebo; Cohort 2-Placebo; Cohort 3-Placebo; Cohort 4- Placebo; Cohort 5- Placebo; Cohort 6- Placebo

SUMMARY:
This is a dose escalation/dose finding, double-blind, placebo-controlled, parallel study of GSK2126458 in subjects with IPF. The study is designed to explore a number of doses of GSK2126458 for engagement of pharmacology after short term dosing. It is anticipated that approximately 24 subjects will be enrolled in this study. Actual number of cohorts in this study could vary up to a maximum of 6 cohorts (n=4/cohort; 3 on active and 1 on placebo).

Each cohort will consist of four subjects who will be randomised to receive GSK2126458 (three subjects) or placebo (one subject) for approximately 8 days (7 to 10 days). On Day 1 they will receive their first dose of GSK2126458 (or placebo) and safety, tolerability and PK/PD in the blood will be measured for up to 8 hours post-dose. Subjects will then be discharged from the site with study drug until the last day of dosing. They will also receive hand held spirometers and instructions on action to be taken in case of deterioration in pulmonary function or any other adverse events (AEs). On the last day of dosing they will return to the site for a repeat of the Day 1 procedures.

A bronchoalveolar lavage (BAL) and [18F]-fluoro-deoxyglucose (FDG)- positron emission tomography / computed tomography (PET/CT) scan will be conducted twice during the study; once, at least 2 days before dosing commences and again during the course of the dosing period.

After the final subject in each cohort has completed dosing, a dose escalation meeting will take place. Safety and tolerability and PK data will be reviewed during this meeting and decisions made may include but are not limited to: escalate the dose, decrease the dose or repeat the same dose in the next cohort; stop the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF as determined by a responsible and experienced chest physician and based on established criteria defined by the American Thoracic Society/European Respiratory Society: American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias.
* FVC greater than (>) 40% predicted and Diffusing capacity of the Lung for Carbon Monoxide (DLCO) >30% predicted
* Alanine aminotransferase (ALT) less than (<) 2x upper limit of normal (ULN); alkaline phosphatase and bilirubin less than or equal to (<=) 1.5xULN.
* QTcB <450 milliseconds (msec) and QTc interval <=480 msec; or QTc <480 msec in subjects with Bundle Branch Block.
* Male over 45 years of age inclusive, or female over 50 years of age inclusive at the time of signing the informed consent
* A female subject is eligible to participate if she is of non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhoea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception, if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2 to 4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until the follow-up contact.
* Body weight >=40 kilogram (kg) (female), >=50 kg (male), and body mass index (BMI) between 20 and 35 kg/meter squared (m^2) inclusive.
* Subjects must have left ventricular ejection fraction (LVEF) >=50 % as demonstrated by a recent echocardiogram (at screening or within 3 months prior to screening).

Exclusion Criteria:

* Current IPF exacerbation
* History of acute coronary syndromes, atrial fibrillation, coronary angioplasty, or stenting within the past 24 weeks.
* Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* Uncontrolled hypertension or a history of conditions which could increase the risk of complications from hypertension
* Current upper or lower respiratory tract infection
* Repeated systolic BP >=160 millimeters of mercury (mmHg) and/or diastolic BP >=90 mmHg unless they are diabetic, in which case subjects with repeated systolic BP >=145 mmHg and/or diastolic >=85 mmHg
* Poorly controlled diabetes (HbA1c [glycated hemoglobin (hemoglobin A1c)] >7.5%).
* Clinically significant laboratory assessment outside the reference range unless the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* Previous exposure to ionising radiation >5 millisievert (mSv) in the 3 years prior to enrolment
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (approximately 240 milliliters [mL]) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* Subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Currently taking Pirfenidone or have received Pirfenidone within the previous 30 days
* Unable to refrain from the use of prohibited prescription or non-prescription drugs, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety
* History of sensitivity to any of the study medications, or components there of or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* History of sensitivity to heparin or heparin-induced thrombocytopenia

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-03-08 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic (PD) endpoints pAKT/AKT in platelet-rich plasma and BAL cells, [18F]-FDG-PET/CT | Baseline, Day 1, mid-study BAL visit (Day 5-9) and final dosing day (Day 7, 8, 9 or 10) for each cohort
  Pharmacodynamic will be measured by inhibition of pAKT/AKT in platelet-rich plasma and BAL cells, as well as inhibition of glucose uptake as measured by thoracic[18F]-FDG-PET/CT
Area under the curve (AUC) in blood for GSK2126458 | Day 1, mid-study PET visit (Day 4-8), mid-study BAL visit (Day 5-9) and final dosing day post-dose (Day 7, 8, 9 or 10) for each cohort
  GSK2126458 PK parameters in blood in order to define the blood and pulmonary PK/PD relationship for GSK2126458 in IPF subjects
Maximum observed concentration (Cmax) in blood for GSK2126458 | Day 1, mid-study PET visit (Day 4-8), mid-study BAL visit (Day 5-9) and final dosing day post-dose (Day 7, 8, 9 or 10) for each cohort
  GSK2126458 PK parameters in blood in order to define the blood and pulmonary PK/PD relationship for GSK2126458 in IPF subjects
Pre-dose (trough) concentration at the end of the dosing interval (Ctrough) in blood for GSK2126458 | Day 1, mid-study PET visit (Day 4-8), mid-study BAL visit (Day 5-9) and final dosing day post-dose (Day 7, 8, 9 or 10) for each cohort
  GSK2126458 PK parameters in blood in order to define the blood and pulmonary PK/PD relationship for GSK2126458 in IPF subjects
Concentration of GSK2126458 in bronchoalveolar lavage fluid (BALF) | Baseline BAL visit and mid-study BAL visit (Day 5-9).
  GSK2126458 concentration in BALF in order to define the pulmonary PK/PD relationship for GSK2126458 in IPF subjects

SECONDARY OUTCOMES:
Safety and tolerability of GSK2126458 as assessed by number of subjects with adverse events (AE)s | Baseline up to final dosing day (Day 7, 8, 9 or 10) for each cohort
  Safety and tolerability parameters will include recording of AEs, throughout the study in subjects with IPF
Safety and tolerability of GSK2126458 as assessed by change from baseline in vital signs | Day 1, final dosing day (Day 7, 8, 9 or 10) and follow-up (10-14 days post last dose), for each cohort
  Vital sign measurement will be done in a semi-supine position and will include systolic and diastolic blood pressure, pulse rate and tympanic temperature
Safety and tolerability of GSK2126458 as assessed by change from baseline in clinical laboratory parameters | Day 1, mid-study BAL visit (Day 5-9), final dosing day (Day 7, 8, 9 or 10) and follow-up (10-14 days post last dose) for each cohort
  Clinical laboratory assessments will include haematology, clinical chemistry, urinalysis and additional parameters
Safety and tolerability of GSK2126458 as assessed by change from baseline in pulmonary function | Recorded daily from screening until final dosing day (Day 7, 8, 9 or 10) for each cohort
  Pulmonary function will be assessed by spirometry to test the forced expiratory volume in one second (FEV1) and forced vital capacity (FVC)
Safety and tolerability of GSK2126458 as assessed by change from baseline in electrocardiogram (ECG) | Screening, Day 1 and final dosing day (Day 7, 8, 9 or 10) for each study cohort
  Single 12-lead ECG will be obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTc intervals
Assessment of subject's breathlessness using MRC dyspnoea scale | Day 1 and final dosing day (Day 7, 8, 9 or 10) for each study cohort
  The Medical Research Council (MRC) dyspnoea scale is a 5-point scale used for grading the degree of a patient's breathlessness.
Assessment of FEV1 and FVC using daily hand-held spirometry | Recorded daily from screening until final dosing day (Day 7, 8, 9 or 10) for each cohort
  Subjects will be required to record their daily spirometry scores (FEV1 and FVC) using hand-held spirometers, at approximately the same time each morning between Screening and the Final Dosing Day
Investigate the effect of GSK2126458 on the frequency and or severity of chronic cough using Leicester Cough Questionnaire (LCQ) in IPF subjects | Day 1 and final dosing day (Day 7, 8, 9 or 10) for each cohort
  Subjects will be required to complete the 19 questions - LCQ, which is a symptom specific questionnaire designed to assess the impact of cough severity, a major symptom of IPF. Subjects will be required to complete the 19 questions of the LCQ on Day 1 and the Final Dosing Day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20056

REFERENCES:
- [Background] Lukey PT, Harrison SA, Yang S, Man Y, Holman BF, Rashidnasab A, Azzopardi G, Grayer M, Simpson JK, Bareille P, Paul L, Woodcock HV, Toshner R, Saunders P, Molyneaux PL, Thielemans K, Wilson FJ, Mercer PF, Chambers RC, Groves AM, Fahy WA, Marshall RP, Maher TM. A randomised, placebo-controlled study of omipalisib (PI3K/mTOR) in idiopathic pulmonary fibrosis. Eur Respir J. 2019 Mar 18;53(3):1801992. doi: 10.1183/13993003.01992-2018. Print 2019 Mar. PMID 30765508
- [Derived] Mercer PF, Woodcock HV, Eley JD, Plate M, Sulikowski MG, Durrenberger PF, Franklin L, Nanthakumar CB, Man Y, Genovese F, McAnulty RJ, Yang S, Maher TM, Nicholson AG, Blanchard AD, Marshall RP, Lukey PT, Chambers RC. Exploration of a potent PI3 kinase/mTOR inhibitor as a novel anti-fibrotic agent in IPF. Thorax. 2016 Aug;71(8):701-11. doi: 10.1136/thoraxjnl-2015-207429. Epub 2016 Apr 21. PMID 27103349
- See also: Results for study 116711 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116711?search=study&search_terms=116711#rs